CLINICAL TRIAL: NCT00894673
Title: Randomized Clinical Trial of Sodium Heparin Effectiveness and Security in Patients Submitted to Heart Surgery Using Bypass
Brief Title: Efficacy and Safety of Sodium Heparin (Hipolabor) in Patients
Acronym: HEPSBCCV0109
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Responsible Party: Alexandre Frederico, LAL Clínica Pesquisa e Desenvolvimento Ltda.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HEPSBCCV0109_HIP; (Version 8)
Record Dates: First submitted 2009-05-05; First posted 2009-05-07 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Cardiac Surgery
Keywords: heparin cardiac surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Heparin sodium Hipolabor
  Interventions: Biological: Heparin sodium Hipolabor
- 2 (Active Comparator): Heparim Sodium APP 5.000 USP
  Interventions: Biological: Heparin sodium APP

INTERVENTIONS:
Biological: Heparin sodium Hipolabor — Heparin sodium Hipolabor 5.000 UI/mL
  Arms: 1
Biological: Heparin sodium APP — Heparin sodium APP 5.000 USP
  Arms: 2

SUMMARY:
The objective of this study is to verify, through a randomized, single-blind, multicentre, parallel and comparative study, the effectiveness of heparin sodium of porcine origin in patients undergoing heart surgery at that require the aid of cardiopulmonary bypass, through the control of hemostasis during and after surgery, based on the strengths of markers of coagulation TCA, TTPA, Anti-Xa, heparin bioavailable and loss of excessive blood (bleeding) at the end of the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agree with all aspects of the study and sign the FICT;
* Patients of both sexes;
* Patients aged above 18 years;
* Patients with cardiac surgery and requiring movement; AND
* Extracorporeal.

Exclusion Criteria:

* Patients with hematological disorders that compromise the surgical changes (eg myeloproliferative syndromes, anemia Hb <11.0 g / dL,
* Platelets < 150,000 mm3);
* Patients with disorders of hemostasis (INR> 1.40) (rTTPA> 1.40);
* Patients with renal dysfunction (creatinine> 1.50);
* Patients with deep hyperthermia;
* Liver disease (AST and ALT> 2 times that of the reference value);
* Patients with a history of allergy to heparin or protamine;
* Patients with history of heparin-induced thrombocytopenia;
* Tables infection (eg endocarditis, infection of immune human (HIV), hepatitis B and C, septicemia and pneumonia);
* Reoperations;
* Use of antiplatelet (clopidogrel and ticlopidine) for less than 7 days;
* Use of acetylsalicylic acid is less than 5 days;
* Use of low molecular weight heparin for less than 24 hours; OR
* Use of non-fractioned heparin for less than 12 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2009-07; Primary Completion 2011-07 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Effectiveness of heparin of porcine origin in patients undergoing cardiovascular surgery | 48 hours after surgery.
  Patients undergoing cardiovascular surgery and who require the assistance of cardiopulmonary bypass, through the control of hemostasis during and after surgery, based on measurements of coagulation markers ACT, aPTT, anti-Xa heparin serum and excessive blood loss (hemorrhage ) after the final surgery.

SECONDARY OUTCOMES:
Evaluation of the average dose and and safety of porcine heparin. | 48 hours after surgery.
  Evaluate the mean dose of heparin used in surgery and its relationship to the dose of protamine chloride and the need for blood transfusions and blood products during and after the process

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Lal Clinica Pesquisa e Desenvolvimento Ltda, Valinhos, São Paulo
  - LAL Clinica, Valinhos, São Paulo